CLINICAL TRIAL: NCT03699488
Title: Asynchronous Messaging Therapy for Depression and Anxiety: A Longitudinal Study
Brief Title: Messaging Therapy for Depression and Anxiety: A Longitudinal Effectiveness Study
Status: Completed | Type: Observational
Sponsor: Talkspace (Industry)
Collaborators: Columbia University (Other); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 1001
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Depressive Symptoms; Anxiety Disorders
Keywords: technology; messaging psychotherapy; depression; anxiety; telehealth
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: psychotherapy via asynchronous message — Behavioral psychotherapy delivered by asynchronous message using the Talkspace application

SUMMARY:
Therapies delivered via technology have been developed to improve accessibility, however, there is limited research regarding messaging therapy in particular, and none that we know of utilizing a longitudinal effectiveness design. The aim of this study was to investigate the overall effectiveness of messaging therapy, identify any contributors to its effectiveness, and to evaluate a dosage effect for this type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Depression and/or Anxiety Disorder

Exclusion Criteria:

* Any psychosis related symptoms or disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals seeking psychotherapy services through digitally-mediated application who present with and are diagnosed with a depression and/or anxiety related disorder.
Sampling Method: Probability Sample
Enrollment: 12980 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Depressive symptoms on the Patient Health Questionnaire - 9 | Up to 52 weeks
  Patient Health Questionnaire - 9 (PHQ-9) is a measure of depression symptoms. It has 9 items, with a minimum of 0 and a maximum of 27, with higher scores indicating more symptoms and distress. Decreasing scores indicate better outcome. All items are summed to give the summary score.
Change from Baseline in Anxiety symptoms on the Generalized Anxiety Disorder - 7 | Up to 52 weeks
  Generalized Anxiety Disorder - 7 (GAD-7) is a measure of anxiety symptoms. It has 7 items, with a minimum of 0 and a maximum of 21, with higher scores indicating more symptoms and distress. Decreasing scores indicate better outcome. All items are summed to give the summary score.

SECONDARY OUTCOMES:
Mean number of words sent from patient to therapist | Up to 52 weeks
  Word counts of the words contained within messages sent
Mean number of words sent from therapist to patient | Up to 52 weeks
  Word counts of the words contained within messages sent

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Malgaroli, PhD, Principal Investigator — New York University

IPD SHARING:
Plan to Share IPD: Yes
IPD for both studies is available in addition to the study protocol and statistical analysis plan. IPD includes demographic information for patient and therapist, as well as outcome scale summary scores for each time point.
Supporting Information: SAP
Time Frame: Data is available from October 10, 2018 to October 10, 2019

REFERENCES:
- [Derived] Hull TD, Malgaroli M, Connolly PS, Feuerstein S, Simon NM. Two-way messaging therapy for depression and anxiety: longitudinal response trajectories. BMC Psychiatry. 2020 Jun 12;20(1):297. doi: 10.1186/s12888-020-02721-x. PMID 32532225